CLINICAL TRIAL: NCT02109484
Title: Phase I/II Descending Age Double-blinded Randomized Placebo-controlled Dose Escalation Study to Examine the Safety Reactogenicity Tolerability & Immunogenicity of the P2-VP8 Subunit Parenteral Rotavirus Vaccine in Healthy Toddlers & Infants
Brief Title: Phase I/II Descending Age Study of P2VP8 Subunit Parenteral Rotavirus Vaccine in Healthy Toddlers and Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC-013; NCT02132156 (obsolete NCT alias)
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Evaluation of a Rotavirus Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort A P2-VP8 30 mcg (Experimental): Cohort A toddlers (24-35 mo) receiving P2-VP8 Subunit Vaccine (30 mcg)
  Interventions: Biological: P2-VP8 Subunit Vaccine 30 mcg
- Cohort A Placebo (Placebo Comparator): Cohort A toddlers (24-35 mo)
  Interventions: Other: Placebo
- Cohort A P2-VP8 60 mcg (Experimental): Cohort A toddlers (24-35 mo) receiving high dose P2-VP8 Subunit Vaccine (60mcg)
  Interventions: Biological: P2-VP8 Subunit Vaccine 60mcg
- Cohort B P2-VP8 10mcg (Experimental): Cohort B infants receiving P2-VP8 Subunit Vaccine (10mcg)
  Interventions: Biological: P2-VP8 Subunit Vaccine 10mcg
- Cohort B placebo (Placebo Comparator): Cohort B infants aged 6 to < 8 weeks receiving placebo
  Interventions: Other: Placebo
- Cohort B P2-VP8 30mcg (Experimental): Cohort B infants aged 6 to < 8 weeks receiving P2-VP8 Subunit Vaccine (30mcg)
  Interventions: Biological: P2-VP8 Subunit Vaccine 30 mcg
- Cohort B1 P2-VP8 60mcg (Experimental): Cohort B1 Infants aged 6 to < 8 weeks receiving P2-VP8 Subunit Vaccine (60mcg)
  Interventions: Biological: P2-VP8 Subunit Vaccine 60mcg
- Cohort A P2-VP8 10mcg (Experimental): Cohort A toddlers (24-35 mo) receiving P2VP8 Subunit Vaccine (10mcg)
  Interventions: Biological: P2-VP8 Subunit Vaccine 10mcg

INTERVENTIONS:
Biological: P2-VP8 Subunit Vaccine 10mcg — 10 mcg
  Arms: Cohort A P2-VP8 10mcg; Cohort B P2-VP8 10mcg
Biological: P2-VP8 Subunit Vaccine 30 mcg — 30 mcg
  Arms: Cohort A P2-VP8 30 mcg; Cohort B P2-VP8 30mcg
Biological: P2-VP8 Subunit Vaccine 60mcg — 60 mcg
  Arms: Cohort A P2-VP8 60 mcg; Cohort B1 P2-VP8 60mcg
Other: Placebo
  Arms: Cohort A Placebo; Cohort B placebo

SUMMARY:
This is is a study of a parenteral rotavirus vaccine (P2-VP8 subunit rotavirus vaccine). The study will examine the safety and immunogenicity of this vaccine first in healthy South African toddlers. If the safety profile is deemed appropriate, the study will continue to explore the safety and immunogenicity of the vaccine in healthy South African infants.

The primary safety hypothesis is that the P2-VP8 subunit rotavirus vaccine is safe and well-tolerated in healthy toddlers and infants. The primary immunogenicity hypothesis is that the P2-VP8 subunit rotavirus vaccine is immunogenic in infant participants and will induce an immune response in at least 80% of participants in at least one of the study groups.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants/toddlers as established by medical history and clinical examination before entering study
* age:

  * toddler cohort: > or = 2 and <3 years old at the time of enrollment
  * infant cohort: > or = 6 and <8 weeks at the time of enrollment
* parental ability and willingness to provide informed consent
* parental intention to remain in the area with the child during the study period.

Exclusion Criteria:

* Presence of fever on the day of enrollment
* Acute disease at the time of enrollment
* Concurrent participation in another clinical trial throughout the entire timeframe for this study
* Presence of malnutrition or any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination that would compromise the participant's health or is likely to result in nonconformance to the protocol
* For infant cohort, history of premature birth (<37 weeks gestation)
* History of congenital abdominal disorders, intussusception, or abdominal surgery
* Known or suspected impairment of immunological function based on medical history and physical examination
* For infant cohort only, prior receipt of rotavirus vaccine
* A known sensitivity or allergy to any components of the study vaccine
* History of anaphylactic reaction
* Major congenital or genetic defect
* Participant's parents not able, available or willing to accept active weekly follow-up by the study staff
* Has received any immunoglobulin therapy and/or blood products since birth or planned administration during the study period
* History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including corticosteroids. Infants on inhaled or topical steroids may be permitted to participate in the study
* Any medical condition in the parents/infant that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parents' ability to give informed consent
* HIV infection

  * For toddlers, to be assessed by HIV ELISA
  * For infants, to be assessed by PCR, if mother is not known to be negative (negative test result between 24 weeks gestation and screening)

Ages: 6 Weeks to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 204 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Groome, Principal Investigator — SAMRC Respiratory and Meningeal Pathogen Research Unit
Locations (1):
- Respiratory and Meningeal Pathogens Research Unit (RMPRU), Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koen A, Jose L, Madhi SA, Fix A, Cryz S, Groome MJ. Neutrophil Counts in Healthy South African Infants: Implications for Enrollment and Adverse Event Grading in Clinical Trials in an African Setting. J Pediatr X. 2019 Spring;1:100005. doi: 10.1016/j.ympdx.2019.100005. PMID 32734176
- [Derived] Groome MJ, Koen A, Fix A, Page N, Jose L, Madhi SA, McNeal M, Dally L, Cho I, Power M, Flores J, Cryz S. Safety and immunogenicity of a parenteral P2-VP8-P[8] subunit rotavirus vaccine in toddlers and infants in South Africa: a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2017 Aug;17(8):843-853. doi: 10.1016/S1473-3099(17)30242-6. Epub 2017 May 5. PMID 28483414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Age de-escalation, dose-escalation study enrolling healthy toddlers and infants between 17 March and 29 September 2014 at a single site in South Africa.
Groups:
- Cohort A Placebo: Healthy toddlers aged 2 to <3 months receiving placebo
- Cohort A 10 mcg P2-VP8: Healthy toddlers 2 to <3 yrs of age receiving low dose P2-VP8
- Cohort A 30 mcg P2-VP8: Healthy toddlers aged 2 to <3 yrs receiving an intermediate dose of P2-VP8
- Cohort A 60 mcg P2-VP8: Healthy toddlers aged 2 to < 3 yrs receiving high dose P2-PV8
- Cohort B Placebo: Healthy Infants aged 6 to <8 weeks receiving placebo
- Cohort B 10 mcg P2-VP8: Healthy Infants aged 6 to <8 weeks receiving low dose P2-VP8
- Cohort B 30 mcg P2-VP8: Healthy Infants aged 6 to <8 weeks of age receiving a medium dose of P2-VP8
- Cohort B 60 mcg P2-VP8: Healthy Infants aged 6 to <8 weeks receiving high dose of P2-VP8
Period: Overall Study
Arm/Group | Cohort A Placebo | Cohort A 10 mcg P2-VP8 | Cohort A 30 mcg P2-VP8 | Cohort A 60 mcg P2-VP8 | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Started | 5 | 13 | 12 | 12 | 50 | 12 | 50 | 50
Completed | 5 | 13 | 12 | 11 | 46 | 11 | 47 | 47
Not Completed | 0 | 0 | 0 | 1 | 4 | 1 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Moved away from study area | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A Placebo: Healthy toddlers aged 2 to < 3 years receiving placebo
- Cohort A 10 mcg P2-VP8: Healthy toddlers aged 2 to < 3 years receiving low dose P2-VP8
- Cohort A 30 mcg P2-VP8: Healthy toddlers aged 2 to < 3 years receiving Medium Dose Ps-VP9
- Cohort A 60 mcg P2-VP8: Healthy toddlers aged 2 to < 3 years receiving High Dose P2-VP8
- Cohort B Placebo: Healthy Infants aged 6 to <8 weeks receiving placeblo
- Cohort B 30 mcg P2-VP8: Healthy Infants aged 6 to <8 weeks receiving Medium Dose P2-VP8
- Cohort B 60 mcg P2-VP8: Healthy Infants aged 6 to <8 weeks receiving High Dose P2-VP8
- Total: Total of all reporting groups
Arm/Group | Cohort A Placebo | Cohort A 10 mcg P2-VP8 | Cohort A 30 mcg P2-VP8 | Cohort A 60 mcg P2-VP8 | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8 | Total
Number analyzed (Participants) | 5 | 13 | 12 | 12 | 50 | 12 | 50 | 50 | 204
Age, Continuous [Mean (Full Range); unit: weeks] | 136.4 [126 to 143] | 135.6 [122 to 143] | 139.0 [126 to 152] | 144.7 [139 to 152] | 6.6 [6.1 to 7.7] | 6.6 [6.3 to 7.0] | 6.6 [6.1 to 7.7] | 6.7 [6.1 to 8] | 72.8 [6.1 to 152]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 7 | 6 | 24 | 5 | 23 | 25 | 99
  Male | 2 | 7 | 5 | 6 | 26 | 7 | 27 | 25 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 12 | 12 | 12 | 50 | 12 | 49 | 50 | 202
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 5 | 13 | 12 | 12 | 50 | 12 | 50 | 50 | 204

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaccine Induced Reactions
Description: Maximum severity of all local reactions or systemic reactogenicity after any vaccination
Time Frame: 7 days following each dose
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A 10 mcg P2-VP8: Healthy toddlers aged 2 to <3 months receiving low dose P2-VP8
- Cohort A 30 mcg P2-VP8: Healthy toddlers aged 2 to <3 months receiving Medium Dose P2-VP8
- Cohort A 60 mcg P2-VP8: Healthy toddlers aged 2 to <3 months receiving placebo High Dose P2-VP8
- Cohort B 10 mcg P2-VP8: Healthy infants aged 6 to < 8 weeks receiving Low Dose P2-VP8
Arm/Group | Cohort A Placebo | Cohort A 10 mcg P2-VP8 | Cohort A 30 mcg P2-VP8 | Cohort A 60 mcg P2-VP8 | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Number analyzed (Participants) | 5 | 13 | 12 | 12 | 50 | 12 | 50 | 50
Participants
  None | 3 | 8 | 4 | 6 | 6 | 2 | 5 | 6
  Mild | 1 | 4 | 7 | 5 | 29 | 10 | 35 | 37
  Moderate | 1 | 1 | 1 | 1 | 14 | 0 | 9 | 6
  Severe | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants experiencing a Serious Adverse Event within 28 days of a vaccination and at any time during the study
Time Frame: within 28 days of a study dose and at any time
Population: All subjects that received at least one dose of P2-VP8 vaccine or placebo
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A Placebo: Healthy toddlers aged 2 to <3 years receiving Placebo
- Cohort A 10 mcg P2-VP8: Healthy toddlers aged 2 to <3 years receiving Low Dose P2-VP8
- Cohort A 30 mcg P2-VP8: Healthy toddlers aged 2 to <3 years receiving Medium Dose P2-VP8
- Cohort A 60 mcg P2-VP8: Healthy toddlers aged 2 to <3 years receiving High Dose P2-VP8
Arm/Group | Cohort A Placebo | Cohort A 10 mcg P2-VP8 | Cohort A 30 mcg P2-VP8 | Cohort A 60 mcg P2-VP8 | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Number analyzed (Participants) | 5 | 13 | 12 | 12 | 50 | 12 | 50 | 50
Participants
  SAE within 28 days of vaccine receipt | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 5
  SAE at any time during follow-up | 0 | 0 | 0 | 0 | 4 | 0 | 6 | 6

3. Primary Outcome: Number of Participants Reporting Any Non-Serious Adverse Event
Description: all adverse events will be recorded over the duration of the 6 month follow up period.
Time Frame: 6 mo following first vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A 10 mcg P2-VP8: Healthy toddlers aged 2 to <3 months receiving Low Dose Toddlers P2-VP8
- Cohort A 60 mcg P2-VP8: Healthy toddlers aged 2 to <3 months receiving High Dose P2-VP8
- Cohort B 60 mcg P2-VP8: Healthy Infants aged 6 to <8 weeks receiving High Dose Infants P2-VP8
Arm/Group | Cohort A Placebo | Cohort A 10 mcg P2-VP8 | Cohort A 30 mcg P2-VP8 | Cohort A 60 mcg P2-VP8 | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Number analyzed (Participants) | 5 | 13 | 12 | 12 | 50 | 12 | 50 | 50
Participants | 2 | 7 | 6 | 8 | 41 | 11 | 46 | 42

4. Primary Outcome: Number/Percentage of Infant Participants With Anti-P2-VP8 IgA to P[8] Seroresponse.
Description: Seroresponse is defined as 4 fold rise in Geometric Mean Titer (GMT) between pre-(baseline) and post vaccination (4 weeks after third vaccination). Confidence intervals are displayed as percentages.
Time Frame: Baseline to day 84
Population: Enrolled infants who received 3 vaccinations and with pre and post-vaccination immunologic parameters measured
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Number analyzed (Participants) | 45 | 12 | 47 | 47
Participants | 9 | 7 | 38 | 32
Statistical Analysis 1: Comparison: Cohort B Placebo vs Cohort B 10 mcg P2-VP8; Test type: Equivalence — Power to detect difference between treatment groups for seroresponse between 50% and 95% for P2-VP8 subunit rotiarivus vaccine calculated based on estimate of 10% loss. 45 evaluable participants in 2 highest doses tolerated in B1 infant cohort, study idesigned to provide >= 89% and >= 77% power to detect 35 and 30 percentage points difference, respectively, between the two dose levels and provide > 95% to detect >= 40 percentage point difference between a P2-VP8 dose group and placebo group; p = 0.0165, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort B Placebo vs Cohort B 30 mcg P2-VP8; Power to detect difference between treatment groups for seroresponse between 50% and 95% for P2-VP8 subunit rotiarivus vaccine calculated based on estimate of 10% loss. 45 evaluable participants in 2 highest doses tolerated in B1 infant cohort, study idesigned to provide >= 89% and >= 77% power to detect 35 and 30 percentage points difference, respectively, between the two dose levels and provide > 95% to detect >= 40 percentage point difference between a P2-VP8 dose group and placebo group; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort B Placebo vs Cohort B 60 mcg P2-VP8; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Number/Percentage of Infants With Anti-P2-VP8 IgG to P[8] Seroresponses
Description: Seroresponse is defined as 4 fold rise in Geometric Mean Titer (GMT) between pre-(baseline) and post vaccination (4 weeks after third injection).An unadjusted serioresponse was defined as an increase of 4 times or more in titers between baseline and 4 weeks after the 3rd injection. Adjusted IgG and neutralizing antibody post injection titres accounted for the decay in maternal antibodies using the half-life calculated from participants in the placebo group with detectable baseline titers higher than those at the post injection visit.
Time Frame: Baseline to day 84
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B 30 mcg P2-VP8: Healthy Infants aged 6 to <8 weeks receiving Medium Dose P2-VP8 Medium Dose Infants
Arm/Group | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Number analyzed (Participants) | 45 | 12 | 47 | 47
Participants
  Unadjusted Seroresponse | 1 | 12 | 46 | 46
  Adjusted Seroresponse | 4 | 12 | 46 | 47
Statistical Analysis 1: Comparison: Cohort B Placebo vs Cohort B 30 mcg P2-VP8; Pair-wise comparisons between Cohort B Placebo group and the active vaccination groups were peformed; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort B Placebo vs Cohort B 60 mcg P2-VP8; Test type: Equivalence — Pair-wise comparisons between Cohort B Placebo group and the active vaccination groups were performed; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort B Placebo vs Cohort B 10 mcg P2-VP8; Test type: Equivalence — Pair-wise comparisons between Cohort B Placebo group and the active vaccination groups were performed; p = 0.0006, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Number/Percentage of Infants With Neutralizing Antibody Response to WA Strain (G1[P8])
Description: as for outcome 5
Time Frame: Baseline to Day 84
Population: Enrolled infants who received placebo, 10 mcg, 30 mcg or 60 mcg V2-VP8.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Number analyzed (Participants) | 45 | 12 | 47 | 47
Participants
  Unadjusted seroresponse to neutralizing antibodies | 0 | 7 | 17 | 7
  Adjusted seroresponse to neutralizing antibodies | 3 | 12 | 40 | 40
Statistical Analysis 1: Comparison: Cohort B Placebo vs Cohort B 10 mcg P2-VP8; A pair wise comparison between the Adjusted Seroresponses in the placebo group and the Group B 10 mcg P2-VP8 was performed; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.0004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cohort B Placebo vs Cohort B 30 mcg P2-VP8; A pair wise comparison between the Adjusted Seroresponses in the placebo group and the Cohort B 30 mcg P2-VP8 vaccine group was performed; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cohort B Placebo vs Cohort B 60 mcg P2-VP8; A pair-wise comparison between the Adjusted Seroresponses in Cohort B Placebo group and the Cohort B P2-VP8 group was performed; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.0001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Rotavirus Shedding After Administration of Rotarix in Infants Receiving 3 Doses of Vaccine or Placebo.
Description: Percent of infants who shed rotavirus at any timepoint after receiving 3 doses of study vaccine and one dose of Rotarix. Infants received Rotarix vaccination beginning on Day 84. Stool specimens were collected from these infants on the 5th, 7th and 9th day following first administration of Rotarix. This test was performed as a novel functional assessment of the ability to suppress local gut multiplication of the vaccine strain contained in Rotarix.
Time Frame: Rotarix vaccination on Day 84 to day 91
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B Placebo | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
Number analyzed (Participants) | 44 | 45 | 46
Participants
  Any Timepoint - Rotavirus shedding | 17 | 6 | 9
  No shedding of rotavirus | 27 | 39 | 37

ADVERSE EVENTS:
Time Frame: 28 days after any vaccination
Arm/Group | Cohort A Placebo | Cohort A 10 mcg P2-VP8 | Cohort A 30 mcg P2-VP8 | Cohort A 60 mcg P2-VP8 | Cohort B Placebo | Cohort B 10 mcg P2-VP8 | Cohort B 30 mcg P2-VP8 | Cohort B 60 mcg P2-VP8
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/13 | 0/12 | 0/12 | 0/50 | 0/12 | 0/50 | 2/50
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/13 | 0/12 | 0/12 | 4/50 | 0/12 | 7/50 | 8/50
Other Adverse Events (participants affected / at risk) | 2/5 | 7/13 | 6/12 | 8/12 | 41/50 | 11/12 | 46/50 | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Placebo (N=5) | Cohort A 10 mcg P2-VP8 (N=13) | Cohort A 30 mcg P2-VP8 (N=12) | Cohort A 60 mcg P2-VP8 (N=12) | Cohort B Placebo (N=50) | Cohort B 10 mcg P2-VP8 (N=12) | Cohort B 30 mcg P2-VP8 (N=50) | Cohort B 60 mcg P2-VP8 (N=50)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Acute gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Death unknown cause
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Placebo (N=5) | Cohort A 10 mcg P2-VP8 (N=13) | Cohort A 30 mcg P2-VP8 (N=12) | Cohort A 60 mcg P2-VP8 (N=12) | Cohort B Placebo (N=50) | Cohort B 10 mcg P2-VP8 (N=12) | Cohort B 30 mcg P2-VP8 (N=50) | Cohort B 60 mcg P2-VP8 (N=50)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 8 (8) | 6 (8)
Candida nappy rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Conjuntivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 5 (5) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 4 (4) | 3 (3)
Helminthic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 24 (31) | 5 (6) | 25 (31) | 30 (40)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 3 (3) | 6 (6) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 15 (16) | 2 (2) | 14 (15) | 7 (8)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dermatitiis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 5 (5) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 2 (2) | 2 (2) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No